CLINICAL TRIAL: NCT02872493
Title: Observational Study of the Effect of Small Intestine Length on Bariatric Surgical Patient Outcomes
Brief Title: Small Bowel Length and Bariatric Surgery Outcomes
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Charles R. Flynn, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: 160971
Record Dates: First submitted 2016-08-08; First posted 2016-08-19 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Malnutrition; Obesity; Weight Loss; Micronutrient Deficiency
Keywords: obesity; bariatric surgery; bowel length
MeSH Terms: conditions — Malnutrition; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RYGB: Roux-en-Y Gastric Bypass - these are patients that undergo a Roux-en-Y gastric bypass operation for their bariatric operation.
  Interventions: Procedure: Small bowel length measurement
- VSG: Vertical Sleeve Gastrectomy - these are patients that undergo a vertical sleeve gastrectomy operation for their bariatric operation.
  Interventions: Procedure: Small bowel length measurement

INTERVENTIONS:
Procedure: Small bowel length measurement — The total length of the small bowel with be measured at the time of the bariatric surgical operation.

SUMMARY:
The purpose of this study is to determine whether or not the total length of small intestine effects outcomes after bariatric surgery in a cohort of patients preoperatively and up to ten years postoperatively. Roux-en-Y gastric bypass and vertical sleeve gastrectomy will be the surgical groups in this study. We aim to determine if bowel length has a significant effect on long term weight loss or other nutritional deficiencies in this bariatric cohort.

DETAILED DESCRIPTION:
Bariatric surgery (also known as "weight loss surgery") is the most effective treatment for obesity as well as a number of other obesity-related conditions, including type 2 diabetes, hypertension, and hypercholesterolemia. Interestingly, not all patients respond with significant weight loss following surgery and some patients even lack much weight loss at all over the long-term. Even though variability in treatment response is observed in a variety of diseases, the biological basis for this variability in weight loss after bariatric surgery is poorly understood. Recent data from our group as well as others, however, suggest that differences in the total length of the small intestine may significantly contribute to these differences in weight loss over time. For example, Roux-en-Y gastric bypass is thought to exert its weight loss effect because of a bypass of small intestine that causes a degree of nutrient malabsorption. The bypassed small intestine (<100cm) is near the proximal end of the intestines closest to the stomach. Hypothetically, an individual with the greater total small intestine length may not benefit as much from the bypass as someone who has a much shorter length of total small intestine. Whether or not this hypothetical relationship is true remains unknown, but a recent study demonstrated that small intestine length does differ significantly between individuals with lengths ranging from 300cm to >1200cm. The total length of small intestine is not routinely measured during any bariatric procedure, as the lengths of the bypass limbs are determined from the portion of the intestines closest to the stomach. The purpose of this study is to determine whether the amount of total small intestine significantly affects weight loss in patients undergoing bariatric surgery - both the Roux-en-Y gastric bypass (RYGB) or the Vertical Sleeve Gastrectomy (VSG). If there is a significant effect of total small intestine length on long-term weight loss in bariatric patients, then it would justify the conduct of a further study to determine whether or not these operations should be performed differently in individuals to account for the differences in small intestine length. This is an observational study that will be looking at body weight (primary endpoint) and other nutritional endpoints (other pre-specified outcome measure) over time up to ten years in this patient cohort. The body weight measurements and any laboratory data will be collected that are part of the routine clinical care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic bariatric surgery, either vertical sleeve gastrectomy or Roux-en-Y gastric bypass
* Able to give informed consent

Exclusion Criteria:

* Prior small intestine resection.
* Inability to safely obtain total small intestinal length measurements in the operating room.
* Any small bowel tethering due to intestinal adhesions identified in the operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be studying two cohorts of patients prior to and following either Roux-en-Y gastric bypass or vertical sleeve gastrectomy for up to ten years.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2016-08; Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Body Weight | Up to 10 years postoperatively as measured for routine clinical care
  Body weight will be measured preoperatively (within 30 days of the operation) as the baseline body weight, then postoperatively up to ten years from the time of initial surgery. Measurements will be made per routine clinical care and not solely for research purposes. Exact time points before and after surgery that body weight will be measured, except for the day of surgery, will differ between patients in the study.
  Change in body weight over time will be measured annually, adjusted for baseline body weight at the time of surgery.
  Regression will be used to test for a significant interaction of "total bowel length" and "body weight" over time in the patient cohorts (RYGB vs. VSG) - this is our primary outcome measurement. We are examining whether there is a significant interaction between any change in body weight over time and the small bowel length in the patient cohorts.

OTHER OUTCOMES:
Vitamin A | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin D | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin E | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin B1 | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin B2 | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin B6 | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Vitamin B12 | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Iron | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Parathyroid Hormone | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Total Iron Binding Capacity | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.
Ferritin | Up to 10 years postoperatively
  Other pre-specified outcomes will be analyzed annually, adjusted for baseline measurements. Similar to the primary endpoint, data will be analyzed as continuous variables and tested for an interaction between total bowel length and the nutritional variable of interest. These other nutritional outcomes will vary depending on the clinical course of the individual patients in this observational study. Thus, time points that patients will have these variables measured will not be exactly the same across patients and will depend on the clinical care of the individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Flynn, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Albaugh VL, Weinberg JL, Yu D, Spann MD, Williams DB, Samuels JM, Flynn CR, English WJ. Total Alimentary Limb Length Is Not Associated with Weight Loss Following Proximal Roux-en-Y Gastric Bypass. Obes Surg. 2025 May;35(5):1693-1701. doi: 10.1007/s11695-025-07817-5. Epub 2025 Mar 27. PMID 40146457
- See also: Total Alimentary Limb Length Is Not Associated with Weight Loss Following Proximal Roux-en-Y Gastric Bypass — https://link.springer.com/article/10.1007/s11695-025-07817-5